CLINICAL TRIAL: NCT06442007
Title: A 3-arm Multi-Center Exploratory Trial of Universally Delivered Interventions for Prevention of Anxiety and Depression in Young People in Pakistan
Brief Title: Universally Delivered Interventions for Young People
Acronym: Mindset-PK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Fatima Jinnah Women University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mindset-PK
Record Dates: First submitted 2024-05-17; First posted 2024-06-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Distress, Emotional
Keywords: adolescents; anxiety; depression; single session interventions; growth mindset; Pakistan
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Three arm study. Schools would be the unit of cluster.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Behavioral Activation - single session intervention (BA-SSI) (Experimental): This is comprised of 5 five components:
  1. Discussion on the rationale of the behavioral activation
  2. Awareness raising about distress, including how behavior shapes feelings and thoughts;
  3. a life values assessment
  4. the creation of an activity action plan
  5. an exercise in which youths write about benefits that might result from engaging in each activity, an obstacle that might keep them from doing the activities and a strategy for overcoming the identified obstacles.
  Interventions: Behavioral: Behavioral Activation - single session intervention (BA-SSI)
- 4-session Mindset intervention (Active Comparator): This is comprised of a growth mindset module (2 sessions), a gratitude module (1 session) and a value affirmations module (1 session). Sessions are delivered weekly (over 4 weeks) and each session lasts for an hour. Reading and writing activities and group discussions are included in each session. Participants are supposed to complete homework exercises are assigned between sessions.
  Interventions: Behavioral: 4-session Mindset intervention
- Waiting list control group (No Intervention): At end of the study, this group will be offered to choose one intervention from two active interventions mentioned above.

INTERVENTIONS:
Behavioral: Behavioral Activation - single session intervention (BA-SSI) — Single session intervention
  Arms: Behavioral Activation - single session intervention (BA-SSI)
Behavioral: 4-session Mindset intervention — This is comprised of 4 sessions.
  Arms: 4-session Mindset intervention

SUMMARY:
Mental health problems are amongst the major contributors to disease burden globally.

According to a recent study, 34% of young people worldwide (aged 10-19) suffer from depression and more than half of this population belongs to Southeast Asia such as Pakistan, India, and China.

Existing evidence shows that the access to mental health services in LMICs is limited and even fewer child psychiatric services are available.

One approach to overcome barriers such as limited availability of trained mental health professionals and risk of stigma may involve the use of simple, brief, scalable interventions based on basic psychological principles rather than treatment of psychopathology.

This study adapts and evaluates two brief interventions called behavioral activation single session intervention (BA-SSI) and 4-session Mindset intervention (MI) for teenage depression and anxiety in Pakistan, where access to mental health care is constrained by societal stigma and a shortage of clinicians.

DETAILED DESCRIPTION:
A 3-arm multi-center cluster exploratory Randomized Controlled Trial to determine the feasibility, acceptability and preliminary effectiveness of a universally delivered, culturally adapted, potentially low cost, 4-session Mindset intervention (MI) and behavioral activation single session intervention (BA-SSI) for school going young persons (YP) (12-15 years) in Pakistan.

Proposed study is designed using the updated Medical Research Council (MRC) Framework for the development and evaluation of complex interventions.

Three public schools will be recruited from each of 10 cities across Pakistan: Karachi, Hyderabad, Nawabshah, Thatta, Lahore, Gujrat, Rawalpindi, Multan, Quetta, and Peshawar.

All the participants, regardless of their treatment arm, will be assessed at baseline, 1 month post-baseline and at 3-month.

ELIGIBILITY:
Young persons (YP)

Inclusion Criteria:

* Youth is between the age 12-15 years (inclusive) at the time of study enrollment.
* Youth has one parent or legal guardian to give consent.
* Youth speaks Urdu well enough to complete the paper based intervention.

Exclusion Criteria:

* Intellectual disability, as this may undermine comprehension of intervention material.
* Adolescent with history of hospitalization or those who received inpatient treatment for a mental health problem within the past two months as the intervention being tested and this study is not designed for adolescent with acute medical and/or psychiatric treatment needs (if identified with any acute medical and/or psychiatric problem, they would be referred to appropriate health services through parents).

Schools Inclusion Criteria

Schools in the study areas are eligible to participate if they meet all the following criteria:

1. the school authority agrees to participate;
2. the schools shall be non-specialist public schools;
3. school contains at least 80 students; Exclusion criteria

If the school meet the following exclusion criteria, they are ineligible to participate:

1. the school authority refuses to participate;
2. a specialist and/or independent or private school;

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 564 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Total recruitment period is 3 months. Change in numbers will be recorded from first month of recruitment to 3rd month of recruitment
  This will be monitored through a research trial log. This log will include information about number of schools approached, number of schools eligible to participate, number of schools consented to participate, number of YP approached, number of eligible YP and number of those who consented to participate
Feasibility of intervention | Retention of participants in the Intervention at the completion of one month intervention period.
  Session attendance for each participant in active study arms for each session will be recorded and maintained in participant intervention log.
Depression | Change in scores from baseline to 3-month follow up.
  The Patient Health Questionnaire -8 will be used to assess the symptoms of depression. PHQ-8 scores are highly correlated with PHQ-9 scores, and the same cutoffs can be used to assess depression severity

SECONDARY OUTCOMES:
The Revised Child Anxiety and Depression Scale | Change in scores from baseline to 3-month follow up
  It is a 47-item, youth self-report questionnaire with subscales including: separation anxiety disorder (SAD), social phobia (SP), generalized anxiety disorder (GAD), panic disorder (PD), obsessive compulsive disorder (OCD), and major depressive disorder (MDD). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). Items are rated on a 4-point Likert-scale from 0 ("never") to 3 ("always").
Growth Mindset scale | Change in scores from baseline to 3-month follow up
  The mindset scale is comprised of 3 items regarding participants' views about the mindset such as intelligence, personality etc. There is not cutoff score. Higher total summed scores indicate stronger ﬁxed mindsets, and lower scores, stronger growth mindsets.
Beck's hopelessness Scale short version | Change in scores from baseline to 3-month follow up
  A 4-item short version of the Hopelessness Scale includes all the affective, cognitive and motivational components of hopelessness.
EuroQol Quality of Life scale | Change in scores from baseline to 3-month follow up
  This scale provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys. higher score indicare greater disability. there is no cutoff score.
Program Feedback Scale | Total acceptability score at completion of one month intervention period.
  youths will be asked to complete a series of questions regarding their experience with the intervention to which they were assigned. highre score will indicate greater level of acceptability. there is no cut off score.

CONTACTS AND LOCATIONS:
Locations (1):
- Public school for boys 1, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
This is the feasibility study and interventions will continue to refine and adapt. The IP is owned by the Pakistan Institute of Living and Learning